CLINICAL TRIAL: NCT05290389
Title: Enhancing Strategic Management of Acute Reperfusion and Therapies in Acute Myocardial Infarction Using a Novel Smartphone APPlication (SMART-AMI APP)
Brief Title: A Smartphone APPlication for the Transmission of ECGs in the Management of Patients Presenting With Suspected Heart Attacks in the Hamilton, Niagara, Haldimand, and Brant Area
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Centre for Evidence-Based Implementation (Unknown)
Responsible Party: Sponsor
Other Study IDs: HAH-21-015
Record Dates: First submitted 2022-02-22; First posted 2022-03-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction; STEMI
Keywords: Mixed-methods; Promote Efficient Delivery of Health Care Resources; Technology; Health Care Delivery
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: All Emergency Medicine physicians and Interventional Cardiologists involved in STEMI care in the Hamilton Niagara Haldimand Brant Local Health area will be eligible for participation in this study.
  Interventions: Other: SMART AMI APPLICATION

INTERVENTIONS:
Other: SMART AMI APPLICATION — SMART AMI allows real-time sharing and review of patient history and ECG between Emergency Department physicians and Interventional Cardiologists to allow for immediate decision-making regarding the need for percutaneous coronary intervention.
  Participant physicians will use a smartphone application to communicate, transmit the ECG, and activate the STEMI team. This application enables calling and transmission of up to three images of ECGs, which can be reviewed immediately by the Interventional Cardiologist when communicating with the referring physician.

SUMMARY:
The delivery of timely and appropriate care is crucial for patients with heart attacks. Blocked arteries need immediate intervention to restore blood flow. However, the intervention to open the artery is only available in large, regional hospitals. There are only 18 such hospitals across Ontario. Patients with heart attacks in smaller hospitals, where the majority of patients present, require transfer for specialized services. The smartphone application being evaluated in this study is meant to help with communication between doctors to arrange transfer of such patients.

The current model for communication is based on fax machines or non-secure text messages. Additionally, these are not easily accessible for most physicians, so decisions to transfer patients may be based on incomplete information. Unnecessary transfer, treatments, and procedures expose patients and healthcare providers to undue risk.

Smartphone technology is well integrated into clinical practice and widely accessible. The proposed solution being tested is secure and leverages the accessibility of smartphones. Emergency physicians can use this to quickly, securely, and accurately transmit information ensuring faster and appropriate decision making for transfers.

DETAILED DESCRIPTION:
A multi-centre, mixed methods observational study focused on Emergency Department physicians who care for patients presenting to a regional partner hospital in the Hamilton, Niagara, Haldimand, Brant Local Health Integration Network (Canada) with suspected ST-segment Elevation Myocardial Infarction (STEMI). There are approximately 700 STEMI patients per year transferred and treated in the Hamilton General Hospital Cardiac Catheterization Lab. As this study is expected to run over the course of one year, it is anticipated that aggregate patient level data on approximately 700 STEMI patients in the STEMI database will be reviewed.

The study will use a pre-post design to evaluate the implementation and use of a clinical intervention, the SMART AMI App. The study will use quantitative registry data already being collected via the ongoing SMART-AMI project (e.g., STEMI database), utilization of data collected from the SMART AMI App, and quantitative and qualitative survey data from participating physicians. As the intervention in this study is a change in process to improve communication between Emergency Department physicians and Interventional Cardiologists, the study does not directly involve patients and individual patient consent will not be required. No new patient data will be collected for the purposes of this study.

Descriptive quantitative analysis and thematic qualitative analysis of survey results will be conducted. Descriptive and inferential statistics will be used for quantitative data derived from patient charts/registry and physician surveys. Continuous variables will be described using mean ± standard deviation. An interrupted time series analysis will be used to compare trends on time-based quality of care indicators. Categorical variables, such as false activation, will be described as frequencies and compared using a Fisher exact test or chi-square test.

Funding for this study was provided by the Hamilton Academic Health Sciences Organization (HAHSO) #HAH-21-015.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine physicians at hospitals and urgent care centres located in the Hamilton, Niagara and Brant Local Health area:

  * Brantford General Hospital
  * Fort Erie Urgent Care Center
  * Greater Niagara General Hospital
  * Haldimand War Memorial Hospital
  * Hamilton General Hospital
  * Joseph Brant Hospital
  * Juravinski Hospital
  * Main Street West UCC
  * Norfolk General Hospital
  * Port Colborne Urgent Care Center
  * St. Catharines General Hospital
  * St. Joseph's Hospital
  * St. Joseph's Urgent Care Center
  * Welland County General Hospital
  * West Haldimand General Hospital
  * West Lincoln Memorial Hospital
  * Willett Urgent Care Centre

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians:
  Emergency Medicine physicians working at the partner emergency departments and urgent care centres that refer STEMI patients to the cardiac catheterization lab at Hamilton General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Usability | 12 months
  The first primary outcome is usability of the App for Emergency Medicine physicians. This will be measured using electronic surveys and focus groups to identify barriers and facilitators faced when using the App.
Acceptability | 12 months
  The second primary outcome is acceptability of the App for Emergency Medicine physicians. This will be measured using the mHealth App Usability Questionnaire.
Functionality | 12 months
  The third primary outcome will measure functionality of the App for Emergency Medicine physicians. Through electronic surveys, barriers and facilitators faced when using the App will be assessed.

SECONDARY OUTCOMES:
Implementation | 12 months
  The secondary outcome will measure implementation of the App. This will be acquired by the number of Emergency Medicine physicians who signed up for the App and used the App. This measurement will be acquired from Google Data Analytics.
Timing of Care Intervals | 12 months
  Further secondary outcomes include measuring effectiveness of the App through timing of care intervals. This outcome will be acquired from a consecutive sample of patients from the regional STEMI registry. As these data are already collected as part of the ongoing SMART AMI program, no new patient data will need to be collected for the purpose of this study.
False Positive Activation Rates | 12 months
  Effectiveness of the App will be further measured by false positive STEMI activation rates. This outcome will be acquired from a consecutive sample of patients from the regional STEMI registry. As these data are already collected as part of the ongoing SMART AMI program, no new patient data will need to be collected for the purpose of this study.
STEMI Activations via App | 12 months
  Effectiveness will also be measured by the rate of STEMI activations that utilized the App. This outcome will be acquired from a consecutive sample of patients from the regional STEMI registry. As these data are already collected as part of the ongoing SMART AMI program, no new patient data will need to be collected for the purpose of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Madhu K Natarajan, MD, Principal Investigator — Hamilton Health Sciences Corporation; Mathew Mercuri, PhD, Principal Investigator — Hamilton Health Sciences Corporation; Hassan K Mir, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (17):
- Canada (17):
  - Brantford General Hospital, Brantford, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - Haldimand War Memorial Hospital, Dunnville, Ontario
  - Fort Erie Urgent Care Center, Fort Erie, Ontario
  - West Lincoln Memorial Hospital, Grimsby, Ontario
  - West Haldimand General Hospital, Hagersville, Ontario
  - St. Joseph's Urgent Care Center, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Main Street West UCC, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Greater Niagara General Hospital, Niagara Falls, Ontario
  - Willett Urgent Care Centre, Paris, Ontario
  - Port Colborne Urgent Care Center, Port Colborne, Ontario
  - Norfolk General Hospital, Simcoe, Ontario
  - St. Catharines General Hospital, St. Catharines, Ontario
  - Welland County General Hospital, Welland, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mir H, Cullen KJ, Mosleh K, Setrak R, Jolly S, Tsang M, Rutledge G, Ibrahim Q, Welsford M, Mercuri M, Schwalm JD, Natarajan MK. Smartphone App for Prehospital ECG Transmission in ST-Elevation Myocardial Infarction Activation: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2024 Sep 6;13:e55506. doi: 10.2196/55506. PMID 39240681